CLINICAL TRIAL: NCT05982626
Title: Study of 68Ga /131I SGMIB-ZT-199 PET Imaging Targeting HER2-positive in the Diagnosis of Metastatic Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-545
Record Dates: First submitted 2023-07-07; First posted 2023-08-08 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: HER2-positive Breast Cancer
Keywords: Her2-positive; Metastatic breast cancer; Positron-Emission Tomography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga/131I-SGMIB-ZT-199 (Experimental): 68Ga/131I-SGMIB-ZT-199, single dose
  Interventions: Radiation: 68Ga/131I-SGMIB-ZT-199

INTERVENTIONS:
Radiation: 68Ga/131I-SGMIB-ZT-199 — 68Ga-SGMIB-ZT-199: PET imaging; 131I-SGMIB-ZT-199: SPECT imaging.

SUMMARY:
To evaluate the safety, biodistribution, radiation dosimetry, and uptake in tumor lesions of patients with Her2-positive metastatic breast cancer after injection of [131I]/[68Ga]SGMIB-ZT-199.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients.

  1. Women aged between 18 and 75 years old.
  2. Patients with breast cancer confirmed by histological examination or imaging.
  3. HER2 positive diagnosis confirmed by puncture by immunohistochemistry or fluorescence in situ hybridization (HER2 positive is defined as immunohistochemistry result of 3+ (IHC 3+); or immunohistochemistry result of 2+/positive in situ hybridization result (IHC 2+/ISH+)).
  4. Renal function: serum creatinine less than or equal to the upper limit of the normal range; electrocardiogram: no significant abnormalities.
  5. Patients of childbearing age can cooperate with contraception.
  6. Willing and able to cooperate with all items of this study.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. Severe hepatic or renal insufficiency;
  2. Participation in another study protocol or clinical care within the past year that has resulted in radiation exposure exceeding an effective dose of 50 mSv in addition to the radiation exposure expected from participation in this clinical study.
  3. Participation in this study is considered unsuitable by other investigators.
  4. Pregnant women and other groups unsuitable to receive radiation.
  5. Alcohol allergy, etc.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Dosimetry | about 24hours from time of injection
  To confirm biodistribution and absorbed doses of whole body, tumor lesions, and organs from [131I]SGMIB-ZT-199, assessed by PET/SPECT imaging.

SECONDARY OUTCOMES:
Safety Assessment | From administration of [131I]SGMIB-ZT-199 until 1 week after injection
  Incidence and severity of adverse events (AEs) as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided